CLINICAL TRIAL: NCT00662064
Title: Pharmacology and Physiology of the Lower Urinary Tract
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Prof C J Fowler, Prof C H Fry, Dep Uro-Neurology, National Hospital for Neurology and Neurosurgery, London, UK
Other Study IDs: 00/0039
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Urologic Diseases
Keywords: Lower urinary tract; Physiology; Pathology; Immunohistochemistry; Urinary bladder
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bladder biopsies from patients with lower urinary tract dysfunction and from healthy controls
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients with lower urinary tract dysfunction
- 2: Controls with normal lower urinary tract function

SUMMARY:
The function of the lower urinary tract is simple - urine storage and voiding. However, despite this simplicity of function, the control of the lower urinary tract is a rather complex, multilevel process (urothelium, detrusor, peripheral nerves, spinal cord and higher cerebral centres) and the mechanisms involved remain poorly elucidated.

This study is designed to gain a more in depth understanding of the lower urinary tract function. Using bladder biopsies, tissue staining for characteristic markers present on nerves and other cells will be performed. We hypothesize that certain markers are altered in disease and turn back towards the control level of healthy people or patients with successful medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower urinary tract dysfunction
* Controls with normal lower urinary tract function

Exclusion Criteria:

* Age < 18 years old
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with lower urinary tract dysfunction and controls with normal lower urinary tract function
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2002-02; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemistry + PCR of bladder tissue | not specified (storage of biopsies)

CONTACTS AND LOCATIONS:
Overall Officials: Clare J Fowler, FRCP, Principal Investigator — Department of Uro-Neurology, National Hospital for Neurology and Neurosurgery, University College London Hospitals, London, UK; Suzy Elneil, PhD, MRCOG, Principal Investigator — Department of Uro-Neurology, National Hospital for Neurology and Neurosurgery, University College London Hospitals, London, UK
Locations (1):
- Department of Uro-Neurology, The National Hospital for Neurology and Neurosurgery, London, United Kingdom

REFERENCES:
- [Derived] Roosen A, Datta SN, Chowdhury RA, Patel PM, Kalsi V, Elneil S, Dasgupta P, Kessler TM, Khan S, Panicker J, Fry CH, Brandner S, Fowler CJ, Apostolidis A. Suburothelial myofibroblasts in the human overactive bladder and the effect of botulinum neurotoxin type A treatment. Eur Urol. 2009 Jun;55(6):1440-8. doi: 10.1016/j.eururo.2008.11.009. Epub 2008 Nov 18. PMID 19054608